CLINICAL TRIAL: NCT06639347
Title: An Open Label, Multicenter, Phase Ib/Il Study to Evaluate the Safety, Tolerability, and Efficacy of SHR A2102 in Combination With Other Anti-cancer Agents in Patients With Advanced Urothelial Carcinoma
Brief Title: A Trial of SHR-A2102 With Antitumor Therapy in Advanced Urothelial Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-207
Record Dates: First submitted 2024-10-10; First posted 2024-10-15 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-10

CONDITIONS: Advanced Urothelial Carcinoma

STUDY DESIGN:
Intervention Model Description: SHR-A2102 with antitumor therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A2102 + Adebrelimab injection+SHR-8068 injection (Experimental)
  Interventions: Drug: SHR-A2102; Drug: Adebrelimab injection; Drug: SHR-8068 injection

INTERVENTIONS:
Drug: SHR-A2102 — SHR-A2102
Drug: Adebrelimab injection — Adebrelimab injection
Drug: SHR-8068 injection — SHR-8068 injection

SUMMARY:
The study is being conducted to evaluate the safety, tolerability and efficacy of SHR-A2102 for injection with Antitumor Therapy in Advanced Urothelial Carcinoma. To explore the reasonable dosage of SHR-A2102 for Advanced Urothelial Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Competent to comprehend, sign, and date an informed consent form.
2. Male or female subjects must be age 18 or older.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
4. Subjects must have histologically documented, unresectable locally advanced or
5. Histologically confirmed locally advanced or metastatic urothelial cancer.Phase Ib, subjects must have failed, be intolerant or refused the standard treatment; Phase II, subjects must not have received systemic antitumor therapy for locally advanced unresectable or metastatic urothelial carcinoma.
6. An archival tumor tissue sample or a fresh tissue sample should be provided.
7. Subjects must have measurable disease according to RECIST (version 1.1).

Exclusion Criteria:

1. Subjects with not adequately treated, or uncontrollable , or active CNS metastases.
2. Subjects who have previously received TOPO1-based ADCs.
3. Subjects who have received anti-cancer treatment within 4 weeks prior the first dose of study treatment.
4. Subjects who have received radiotherapy within 14 days , or chest radiotherapy > 30Gy within 6 months prior to the first dose of study drug.
5. Subjects with ongoing clinically significant toxicity associated with prior treatment that has not resolved to ≤ Grade 1.
6. Subjects who have received systemic immunosuppressant treatment within 14 days prior the first dose of study treatment.
7. Subjects who have known or suspected interstitial pneumonitis.
8. Phase Ib: Subjects who have had≥ Grade 3 irAEs during the previous treatment with ICIs.
9. Subjects who have any active, known or suspected autoimmune diseases.
10. Subjects who have moderate or severe ascites with clinical symptoms, or uncontrolled or moderate or above pleural effusion, or pericardial effusion.
11. Subjects who have uncontrolled cardiac diseases or cardiac clinical symptoms.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Phase I: RP2D of SHR-A2102 combined with Adebrelimab and SHR-8068 in patients with advanced urothelial cancer | Up to approximately 5 years
Phase I: Incidence and severity of adverse events | Up to approximately 5 years
Phase II: ORR by investigator assessment | Up to approximately 5 years

SECONDARY OUTCOMES:
Phase I: ORR by investigator assessment | Up to approximately 5 years
Phase I: DCR by investigator assessment | Up to approximately 5 years
Phase I: DoR by investigator assessment | Up to approximately 5 years
Phase I: PFS by investigator assessment | Up to approximately 5 years
Phase I: OS by investigator assessment | Up to approximately 5 years
Phase I: Pharmacokinetic parameter for serum concentrations of SHR-A2102 and free toxin | Up to approximately 5 years
Phase I: Anti-SHR-A2102 antibody (ADA) and anti-SHR-A2102 neutralizing antibody (NAb) | Up to approximately 5 years
Phase II: DCR by investigator assessment | Up to approximately 5 years
Phase II: DoR by investigator assessment | Up to approximately 5 years
Phase II: PFS by investigator assessment | Up to approximately 5 years
Phase II: OS by investigator assessment | Up to approximately 5 years
Phase II: Incidence and severity of adverse events | up to 5 years
Phase II: Pharmacokinetic parameter for serum concentrations of SHR-A2102 and free toxin | Up to approximately 5 years
Phase II: Anti-SHR-A2102 antibody (ADA) and anti-SHR-A2102 neutralizing antibody (NAb) | Up to approximately 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided